CLINICAL TRIAL: NCT01812811
Title: Twentyfour Ambulatory Pulse Wave Velocity and Central Augmentation Index in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Regionshospitalet Silkeborg (Other)
Responsible Party: Sponsor
Other Study IDs: 35522
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Type 2 Diabetes
Keywords: pulse wave analysis; pulse wave velocity; Arteriograph24; Ambulatory; diabetes; reproducibility; diurnal variation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The functionality and reproducibility of pulse wave analysis is investigated in 20 type 2 diabetic patients who had two 24 hour measurements performed within one week with the Arteriograph24 equipment.

DETAILED DESCRIPTION:
Arteriograph24 is a new monitor for measuring ambulatory blood pressure and additional performing brachial cuff based on analysis of a suprasystolic pulse wave.

The study aim to test the feasibility of ambulatory pulse wave analysis every twenty minute (the fraction of missed measurements)and the reprodicility of pulse wave velocity and central augmentation index in type 2 diabetic patients. In addition we will explore the relation between diurnal variation of brachial blood pressure, central blood pressure and pulse wave velocity.

20 type 2 diabetic patients will have 24h ambulatory blood pressure performed twice with an interval of one week.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes

Exclusion Criteria:

* Atrial fibrillation

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes patients recruited from out patient clinic
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Fraction of missed pulse wave analysis | Meaured two times with an interval of one week
  Measurements of ambulatory blood pressure and pulse wave analysis is performed every twenty minute. The fraction of missed measurements of pulse wave analysis during day time and night time analysis is the final outcome

SECONDARY OUTCOMES:
Reproducibility of pulse wave analysis parameters | Measured two times with an interval of one week
  Reproducibility of pulse wave velocity, Central systolic blood pressure and central augmentation index for 24 hour, day and night

OTHER OUTCOMES:
Diurnal variation of brachial blood pressure, central blood pressure and pulse wave velocity | Measured two times with an interval of one week
  brachial blood pressure, central blood pressure and pulse wava velocity is measured evrey twenty minutes and averaged for day time and night time. the relative reduction at nioght for the parameters are calculated

CONTACTS AND LOCATIONS:
Overall Officials: Klavs W Hansen, MD, dr.med., Principal Investigator — Medical department, Diagnostic Center, Regional Hospital Silkeborg, Denmark
Locations (1):
- Medical department, Diagnostic Center, Regional Hospital Silkeborg, Silkeborg, Silkeborg, Denmark